CLINICAL TRIAL: NCT02016053
Title: Incidence and Spectrum of Acute Kidney Injury in Cirrhotics and Assessment of New Biomarkers as Early Predictors of Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-AKI-02
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2014-11

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cirrhosis with baseline renal function: 500 patients of cirrhosis with normal baseline renal function will be enrolled.
- Cirrhosis with Acute Kidney Injury (AKI).: Cirrhotics patients who present with AKI (Acute Kidney Injury) will be enrolled.

SUMMARY:
500 patients with normal renal function will be prospectively studied and incidence, spectrum and natural history of AKI (Acute Kidney Injury) will be observed in them and in 200 patients with abnormal renal function fulfilling AKI (Acute Kidney Injury) criteria will be prospectively studied for 1 year. Also biomarkers will be studied and validated as early predictors of AKI (Acute Kidney Injury).

ELIGIBILITY:
Inclusion Criteria:

- Group A: 500 patients of cirrhosis with normal baseline renal function will be enrolled Group B : 200 patients who present with AKI (Acute Kidney Injury) will be enrolled

Exclusion Criteria:

* Age < 18 or > 70 years
* Preexisting Chronic Renal Disease
* Patients with obstructive uropathy.
* Cirrhosis with HCC (HepatoCellular Carcinoma).
* Advanced cardiopulmonary disease
* Pregnancy
* Patients with extrahepatic malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients with normal renal function. 200 patients with abnormal renal function fulfilling AKI (Acute Kidney Injury) criteria will be prospectively studied.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The incidence , spectrum and natural history of Acute Kidney Injury in patients with cirrhosis | 1 Year
  Incidence is defined as No. of AKI (Acute Kidney Injury) patients during the follow up period of 1 year.
  Spectrum is defined as Grading of AKIN (Acute Kidney Injury Network) 1,2,3 in different child status (Child A,Child B and Child C) at the end .
  Natural History is defined as Occurrence of AKI (Acute Kidney Injury) and its recovery during the follow up period of 1 year.

SECONDARY OUTCOMES:
To study predictive value of Cystatin C in comparison to serum creatinine as early predictor of development and outcome of AKI in a cohort of Cirrhotics. | 1 Years
To study predictive value of Cystatin C to determine progression or resolution of Acute Kidney Injury | 1 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India